CLINICAL TRIAL: NCT00342095
Title: Hormonal and Environmental Risk Factors for Developing Systemic Lupus Erythematosus: The Carolina Lupus Study (CLU) and Disease Progression and Activity in the Carolina Lupus Study
Brief Title: Hormonal and Environmental Risk Factors for Developing Systemic Lupus Erythematosus: The Carolina Lupus (CLU) Study
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999997002; OH97-E-N002
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2007-03-07

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Autoimmune Diseases; Estrogen; Silica; Pesticides; Major Histocompatibility Complex; Genetic Susceptibility
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases; Genetic Predisposition to Disease

SUMMARY:
Systemic lupus erythematosus (SLE) is severe, chronic, disabling autoimmune disease that significantly affects health status and quality of life. Since the disease occurs most often in young to middle-aged adults, SLE can also affect work and disability. However, there is currently little information on work-related disability from longitudinal, population-based studies of SLE.

Participants were enrolled into the Carolina Lupus Study between February, 1997 and July 1999. We plan to conduct two telephone contacts with patients and one telephone contact with controls in a follow-up study to be conducted in 2001. The first patient contact will follow an introductory letter that describes the follow-up study. This letter provides participants the opportunity (via a toll-free phone number) to decline further contact about this study. The first patient contact will be a short (5 minute) interview in which we determine their current source of lupus-related medical care, timing of next expected visit, and update contact information. The second contact will involve a 60-minute telephone interview covering medical care utilization, current health status (including a patient-administered measure of lupus activity), work and disability issues, psychosocial attributes (e.g. helplessness, social support, daily stressors including race-related issues), and changes in exposures since the initial interview. We will attempt to schedule the patients' interviews within 3 months before or after the patient sees his or her own physician for SLE-related evaluation or treatment. A short (15 minutes or less) telephone interview will be conducted with controls focusing on current health, work status, and daily stresso.

Ddisease damage will be assessed using the System Lupus international Collaborating Clinics (SLICC)/American College of Rheumatology (ACR) Damage Index, a standardized and validated instrument that is completed by the patient's physician.

We will seek death certificates for patients and controls who have died in order to obtain cause of death information. Next-of-kin information from death certificates will not be used.

This study will allow up to determine the feasibility of obtaining reliable data on disease damage from more than 50 physicians involved in the treatment of patients in the Carolina Lupus Study. This developmental work is a necessary foundation for any additional follow-up studies of the Carolina Lupus Study cohort. We will also be able to examine associations with disability in patients and in controls and to examine the contribution of various factors to the increased disease severity experience by African-American SLE patients.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is severe, chronic, disabling autoimmune disease that significantly affects health status and quality of life. Since the disease occurs most often in young to middle-aged adults, SLE can also affect work and disability. However, there is currently little information on work-related disability from longitudinal, population-based studies of SLE.

Disease damage will be assessed using the System Lupus international Collaborating Clinics (SLICC)/American College of Rheumatology (ACR) Damage Index, a standardized and validated instrument that is completed by the patient's physician.

This study will allow us to determine the feasibility of obtaining reliable data on disease damage from more than 50 physicians involved in the treatment of patients in the Carolina Lupus Study. This developmental work is a necessary foundation for any additional follow-up studies of the Carolina Lupus Study cohort. We will also be able to examine associations with disability in patients and in controls and to examine the contribution of various factors to the increased disease severity experience by African-American SLE patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients were eligible for the study if they met the 1997 revised American College of Rheumatology classification criteria for SLE (32, 33), were diagnosed between January 1, 1995 and July 31, 1999, were 18 years or older at study enrollment, had lived within the study area during at least 6 months of the year prior to diagnosis, and could speak and understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 640
Dates: Start 1996-12-17; Study Completion 2007-03-07

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Medical Center, Raleigh, North Carolina
  - NIEHS, Research Triangle Park, Research Triangle Park, North Carolina
  - Medical University of South Carolina, Columbia, South Carolina